CLINICAL TRIAL: NCT01968317
Title: Megestrol Acetate Plus Metformin to Megestrol Acetate in Patients With Endometrial Atypical Hyperplasia or Early Stage Endometrial Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiaojun Chen (Other)
Collaborators: Fudan University (Other); Shanghai 6th People's Hospital (Other); Zhejiang Cancer Hospital (Other); Shanghai Changning Maternity & Infant Health Hospital (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Chen, Deputy Secretary of the Party committee, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 134119a4500
Record Dates: First submitted 2013-10-16; First posted 2013-10-24 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Endometrial Atypical Hyperplasia; Endometrial Adenocarcinoma
Keywords: Endometrial Atypical Hyperplasia; Endometrial Adenocarcinoma; Conservative Medication
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Megestrol Acetate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Megestrol acetate and metformin (Experimental): Patients will receive metformin 500 mg by mouth third daily and megestrol acetate 160 mg by mouth daily for 3 months.Then an hysteroscope will be used to evaluate the endometrial condition, and the findings will be recorded.
  Interventions: Drug: Megestrol acetate and metformin
- Megestrol acetate (Experimental): Patients will receive megestrol acetate 160 mg by mouth daily for 3 months.Then an hysteroscope will be used to evaluate the endometrial condition, and the findings will be recorded.
  Interventions: Drug: Megestrol acetate

INTERVENTIONS:
Drug: Megestrol acetate and metformin — Patients will receive metformin 500 mg by mouth third daily and megestrol acetate 160 mg by mouth daily for 3 months.
  Other Names: Megestrol acetate: Megace; Metformin: Fortamet, Glucophage
  Arms: Megestrol acetate and metformin
Drug: Megestrol acetate — Patients will receive megestrol acetate 160 mg by mouth daily for 3 months.
  Other Names: Megestrol acetate: Megace
  Arms: Megestrol acetate

SUMMARY:
The purpose of this study is to see if megestrol acetate plus metformin will be more effective in returning the endometrial tissue to a normal state than megestrol acetate alone in patients with endometrial atypical hyperplasia or early stage endometrial adenocarcinoma.

DETAILED DESCRIPTION:
After diagnosed of endometrial atypical hyperplasia(EAH) or type I endometrial cancer(EC) by dilatation and curettage (D&C) or hysteroscopy, patients will be enrolled. Age, waist circumstances, blood pressure, basic history of infertility, blood pressure, serum lipid level and side effects will be collected. Blood tests, including triglycerides, high density lipoprotein-cholesterol, fasting blood glucose, liver and kidney function will be performed before treatment to evacuate their metabolic conditions.

Patients are randomized to 1 of 2 treatment groups. Patients will receive metformin 500 mg by mouth third daily and megestrol acetate 160 mg by mouth daily for 3 months on Arm I. Patients will receive megestrol acetate 160 mg PO daily for 3 months on Arm II. Then an hysteroscope will be used to evaluate the endometrial condition, and the findings will be recorded. For patients with EAH, complete response (CR) is defined as the reversion of endometrial atypical hyperplasia to proliferative or secretory endometrium; partial response (PR) is defined as regression to simple or complex hyperplasia without atypia; no response (NR) is defined as the persistence of the disease; and progressive disease (PD) is defined as the appearance of endometrial cancer in patients. EAH after treatment will be defined as PR in patients with EC. Continuous therapies will be needed in PR, NR or PD.

After completion of study treatment, 3 months of maintenance treatment will be recommended for patients with CR, and they will be followed up for 2 years.

In addition, we've already had a pilot study in 19 patients primarily diagnosed of endometrial atypical hyperplasia from August 2012 to April 2013. 10 patients were in Arm I and 9 patients were in Arm II. Metabolic syndrome were evaluated among all subjects. After treatment, megestrol acetate plus metformin worked better than megestrol acetate alone. But two arms showed no difference in NR patients, which may suggest metformin just worked as an antitumor drug more than an insulin sensitizer. More supportive researches are needed to verify it.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-45 years old
* Primarily have a confirmed diagnosis of endometrial atypical hyperplasia based upon D&C or hysteroscopy

  * OR primarily have a confirmed diagnosis of endometrial adenocarcinoma(G1, low tumor grade), based upon D&C or hysteroscopy, and three MRI parameters shows there's no myometrial invasion, extension beyond corpus, or enlarged lymph nodes
* Have a desire for remaining reproductive function or uterus
* Need to be able to undergo correlative treatment and follow-up

Exclusion Criteria:

* Have a history of serious liver or renal dysfunction
* Have a confirmed diagnosis of malignant tumor in genital system
* Have taken oral contraceptive or other medicine for the treatment of endometrial hyperplasia in the past 6 months
* Ask for removal of the uterus or other conservative treatment
* serum CA-125 > 35 Um/L

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Chen, PhD, Study Chair — Obstetrics & Gynecology Hospital of Fudan University
Locations (5):
- China (5):
  - Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Changning Maternity & Infant Health Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 307 patients from Obstetrics and Gynaecology Hospital of Fudan University (Shanghai, China) were enrolled to this study between October 2013 to October 2017, including 237 patients with atypical endometrial hyperplasia (AEH) and 70 patients with well-differentiated endometrioid endometrial cancer (EEC).
Pre-assignment Details: 157 of 307 enrolled patients were deemed ineligible, including 28 patients with hysterectomy history, 31 patients with AEH/EEC history, 67 patients with progestin use history, 10 patients refusing to attend this trial, 21 patients transferred to other hospital were excluded from this trial.
Period: Overall Study
Arm/Group | Megestrol Acetate and Metformin | Megestrol Acetate
Started | 76 | 74
Completed | 76 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Megestrol Acetate and Metformin | Megestrol Acetate | Total
Number analyzed (Participants) | 76 | 74 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (4.5) | 33.4 (5.2) | 32.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 74 | 150
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 76 | 74 | 150
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 76 | 74 | 150

OUTCOME MEASURES:

1. Primary Outcome: Cumulative CR Rates Within 16 Weeks
Description: The primary objective was to determine whether metformin plus MA would be associated with a higher CR rate at 3 months of treatment compared with MA alone. However, for patients who eventually underwent the first and second hysteroscopies for endometrium evaluation within 16 weeks of the treatment, the cumulative CR rates within 16 weeks (16w-CR) were analysed as first end point instead of the CR rate at 3 months.
  Complete response was defined as the reversion of AEH/EEC to proliferative or secretory endometrium in pathology.
Time Frame: 16 weeks after initial treatment
Population: In MA+metformin group, 9 cases were excluded in primary analysis for 1 asking for surgery and 8 missing hysteroscopic evaluation.
  In MA group, 16 cases were excluded for 1 asking for surgery and 15 missing hysteroscopic evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- Megestrol Acetate and Metformin: Patients will receive metformin 500 mg by mouth three times daily and megestrol acetate 160 mg by mouth daily. Hysteroscopic evaluation was performed every 3 months during the therapy to evaluate the endometrial condition, and the findings will be recorded.
- Megestrol Acetate: Patients will receive megestrol acetate 160 mg by mouth daily. Hysteroscopic evaluation was performed every 3 months during the therapy to evaluate the endometrial condition, and the findings will be recorded.
Arm/Group | Megestrol Acetate and Metformin | Megestrol Acetate
Number analyzed (Participants) | 67 | 58
Participants | 23 | 12

2. Secondary Outcome: Cumulative CR Rates Within 32 Weeks
Description: One of the secondary objectives was between-group comparisons of the cumulative CR rate at 6 months treatment. However, for patients who eventually underwent the second hysteroscopies for endometrium evaluation within 32 weeks of the treatment, the cumulative CR rates within 32 weeks (32w-CR rates) were analysed as secondary end point instead of the CR rate at 6 months.
Time Frame: 32 weeks after initial treatment
Population: In MA+metformin group, 6 cases were excluded in this analysis for 3 asking for surgery and 3 missing hysteroscopic evaluation.
  In MA group, 8 cases were excluded for 2 asking for surgery and 6 missing hysteroscopic evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Megestrol Acetate and Metformin | Megestrol Acetate
Number analyzed (Participants) | 70 | 66
Participants | 52 | 45

3. Secondary Outcome: Recurrence Rate
Description: All patients were followed up till February 2019. Statistics of patients who didn't accept hysterectomy and were not lost to follow up were analyzed.
Time Frame: through study completion, a median time of 33 months
Population: In MA+metformin group, 3 cases were excluded in this analysis for surgery, 3 for lost to follow-up, and 1 for still in treatment.
  In MA group, 2 cases were excluded for surgery and 6 for lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Megestrol Acetate and Metformin | Megestrol Acetate
Number analyzed (Participants) | 69 | 66
Participants | 7 | 6

4. Secondary Outcome: Pregnancy Rate
Description: All patients were followed up till February 2019. The pregnancy rate was calculated only in women who planned for parenthood immediately after achieving CR.
Time Frame: through study completion, a median time of 33 months
Population: In MA+metformin group only 31 cases wanted to have a baby, and that in MA group were 37.
Measure: Count of Participants; unit: Participants
Arm/Group | Megestrol Acetate and Metformin | Megestrol Acetate
Number analyzed (Participants) | 37 | 31
Participants | 19 | 15

ADVERSE EVENTS:
Time Frame: 32 weeks
Groups:
- Megestrol Acetate and Metformin: Patients will receive metformin 500 mg by mouth three times daily and megestrol acetate 160 mg by mouth daily. After initiating the treatment, hysteroscopic evaluation was performed every 3 months during the therapy to evaluate the endometrial condition, and the findings will be recorded.
- Megestrol Acetate: Patients will receive megestrol acetate 160 mg by mouth daily for 3 months.After initiating the treatment, hysteroscopic evaluation was performed every 3 months during the therapy to evaluate the endometrial condition, and the findings will be recorded.
Arm/Group | Megestrol Acetate and Metformin | Megestrol Acetate
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/74
Other Adverse Events (participants affected / at risk) | 47/76 | 46/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Megestrol Acetate and Metformin (N=76) | Megestrol Acetate (N=74)
Weight gain (Endocrine disorders) | 29 (29) | 34 (34)
Diarrhea (Gastrointestinal disorders) | 12 (12) | 3 (3)
Increased nocturnal urine (Renal and urinary disorders) | 15 (15) | 20 (20)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 (10) | 10 (10)
Breast pain OR Abdominal pain (Vascular disorders) | 17 (17) | 20 (20)
Nausea (Gastrointestinal disorders) | 8 (8) | 4 (4)
Uterine hemorrhage (Congenital, familial and genetic disorders) | 6 (6) | 13 (13)
Dizziness (Nervous system disorders) | 7 (7) | 7 (7)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Insomnia (General disorders) | 2 (2) | 3 (3)
Allergic reaction (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5)
Anorexia (General disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT01968317/Prot_SAP_000.pdf